CLINICAL TRIAL: NCT00527462
Title: Mono-Center, Double-Blind, Cross-Over Study to Explore the Effects of Two Hour Inhalation of Ultrafine Carbon Black Particles Versus Filtered Air on Airway Inflammation Induced by Segmental Allergen Challenge in Asthmatics
Brief Title: Study to Explore the Effects of Two Hour Inhalation of Ultrafine Carbon Black Particles on Airway Inflammation in Asthmatics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Prof. Dr. Norbert Krug, Fraunhofer ITEM
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 07/06 UFP-SFB DFG
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Last update posted 2008-04-30 (Estimated); Status verified 2008-04

CONDITIONS: Asthma
Keywords: Asthma GINA 1
MeSH Terms: conditions — Asthma | interventions — Bronchoscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

INTERVENTIONS:
Procedure: Bronchoscopy — bronchoscopy with segmental allergen challenge
Other: Exposure to ultrafine carbon black particles — Exposure to ultrafine carbon black particles for 2 hours

SUMMARY:
The aim of the study is to test the hypothesis that the allergic airway inflammation in asthmatic patients will be enhanced after exposure to ultrafine particles (UFP). In order to test this in a controlled study, the researchers combine controlled exposure to carbon black model UFP with the well-established model of a segmental allergen challenge, which allows the researchers to safely induce circumscript allergic inflammation in the lung in mild asthmatics. The effect of the UFP on allergic inflammation will be controlled by an inhalation of clean air in a randomized, double-blind, crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, aged 18-45 years.
* Women will be considered for inclusion if they are:

  * Not pregnant, as confirmed by a pregnancy test and not nursing.
  * Not of child-bearing capacity (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal, with documented proof of hysterectomy or tubal ligation, or meets clinical criteria for menopause and has been amenorrheal for more than 1 year prior to the screening visit).
  * Of child-bearing capacity and using a highly effective method of contraception during the entire study (vasectomised partner, sexual abstinence [the lifestyle of the female should be such that there is complete abstinence from intercourse two weeks prior to the first dose of study medication until at least 72 hours after treatment], implants, injectables, combined oral contraceptives, hormonal intrauterine devices [IUDs]).
* Physician diagnosis of mild intermittent seasonal asthma
* Non-smokers, or ex-smokers
* Forced expiratory volume in 1 second (FEV1) > 80% of the predicted value
* Positive skin prick test for grass mix at or within 12 months prior to the screening visit
* Able and willing to give written informed consent to take part in the study
* Available to complete all study measurements
* Able to restrain from particle rich atmosphere (e.g. passive cigarette smoke) within 1 week before exposure to UFP or clean air

Exclusion Criteria:

* Infections of the respiratory tract within the last month
* Past or present disease which, as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, endocrine disease or pulmonary disease (including but not confined to chronic bronchitis, emphysema, tuberculosis, bronchiectasis or cystic fibrosis).
* Pathological findings in safety laboratory tests
* Subjects with clinically relevant infection or known ongoing clinically relevant inflammatory process
* Suspected hypersensitivity to any ingredients of the medication involved with bronchoscopy (bronchodilators, sedatives and local anaesthetics)
* Specific immunotherapy (SIT) within two years prior to the study
* Administration of oral, injectable, or dermal corticosteroids according to 9.2
* Neurological or psychiatric disease or history of drug or alcohol abuse which would interfere with the subject's proper completion of the protocol assignment
* Risk of non-compliance with study procedures
* Participation in another clinical trial 30 days prior to enrolment
* Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study.
* Unlikely to comply with the protocol requirements, instructions and study-related restrictions; e.g., language problems, uncooperative attitude, inability to return for follow-up visits, and improbability of completing the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2007-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
difference of the number of total cells in bronchoalveolar lavage resulting in the comparison of allergenic versus control segments | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Krug, Professor, MD, Principal Investigator — Fraunhofer-Institut, Toxikologie und Experimentelle Medizin
Locations (1):
- Fraunhofer-Institut für Toxikologie und Experimentelle Medizin, Hanover, Lower Saxony, Germany

REFERENCES:
- [Derived] Schaumann F, Fromke C, Dijkstra D, Alessandrini F, Windt H, Karg E, Muller M, Winkler C, Braun A, Koch A, Hohlfeld JM, Behrendt H, Schmid O, Koch W, Schulz H, Krug N. Effects of ultrafine particles on the allergic inflammation in the lung of asthmatics: results of a double-blinded randomized cross-over clinical pilot study. Part Fibre Toxicol. 2014 Sep 10;11:39. doi: 10.1186/s12989-014-0039-3. PMID 25204642